CLINICAL TRIAL: NCT06789718
Title: A Direct-to-Consumer, Randomized, Double-blind, Placebo-controlled Study Assessing the Impact of GABA Probiotic Lactiplantibacillus Plantarum Lp815 on Sleep Outcomes in Participants with Self-Reported Sleep Disturbance
Brief Title: Impact of GABA Probiotic Lactiplantibacillus Plantarum Lp815 on Sleep Outcomes in Participants with Self-Reported Sleep Disturbance
Status: Active, not recruiting | Type: Observational
Sponsor: Verb Biotics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: PS12
Record Dates: First submitted 2025-01-15; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Insomnia (moderate)
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Up to 20 participants (10 per study group) will be consented to participate in an optional substudy that involves collection of urine using a neurotransmitter urine-test at home at 7 timepoints during study period (Baseline, Day 9, 12, 14, 21, 35, and 49 during the study product use period).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Study Product: Participants who meet the study eligibility criteria will be randomly assigned to the study product or the placebo group.
  The study product will contain the GABA Probiotic Lactiplantibacillus plantarum Lp815 (5 Billion cfu/dose) and Microcrystalline Methylcellulose.
  Interventions: Dietary Supplement: GABA Probiotic Lactiplantibacillus plantarum Lp815 (5 Billion cfu/dose)
- Placebo: Participants who meet the study eligibility criteria will be randomly assigned to the study product or the placebo group.
  The study placebo will only contain Microcrystalline Methylcellulose.
  Interventions: Other: Placebo
- Optional Sub-Study: Neurotransmitter Urine Test: Participants who meet the study eligibility criteria and who opt-in to the sub-study will be given the Optional Sub-Study Informed Consent Form and be asked to complete neurotransmitter urine tests during baseline, day 2, day 4, day 7, day 14, day 28, and day 42 in parallel with the main study requirements. The cap for entering the sub-study will be 20 participants out of the 150 on a first-come first-serve basis.
  Interventions: Diagnostic Test: Optional Sub-Study: Neurotransmitter Urine Test

INTERVENTIONS:
Dietary Supplement: GABA Probiotic Lactiplantibacillus plantarum Lp815 (5 Billion cfu/dose) — 75 participants will be randomized into the study product group.
  Groups: Study Product
Other: Placebo — 75 participants will be randomized into the placebo group.
  Groups: Placebo
Diagnostic Test: Optional Sub-Study: Neurotransmitter Urine Test — 20 participants who opt-in to the sub-study will provide urine tests during baseline, day 2, day 4, day 7, day 14, day 28, and day 42 while simultaneously participating in the main-study.
  Groups: Optional Sub-Study: Neurotransmitter Urine Test

SUMMARY:
The rationale for this study is to observe differences in sleep outcomes between a consumer-grade probiotic capsule called GABA Probiotic and a placebo control group. Additionally, the study aims to evaluate the impact of the probiotic product on anxiety, gastrointestinal symptoms, sleep quality, daytime alertness, mood, stress, severity of night sweats (if present), and quality of life. In a subset of participants, the study also aims to evaluate how the probiotic affects neurotransmitter levels in the body using an at-home urinary test. A consumer-driven, decentralized observational clinical research study is therefore well-suited for evaluating the impact of this probiotic product in this population.

DETAILED DESCRIPTION:
Gamma-aminobutyric acid (GABA) is a major inhibitory neurotransmitter in the human nervous system, helping to slow down the stimulation of nerve signals in the brain. GABA plays a pivotal role in calming anxiety, reducing stress and improving sleep. Deficits in GABA levels can lead to a cascade of disorders ranging from anxiety and stress to mood swings and depression. Advancements in understanding the role of the microbiome in the Gut-Brain Axis have highlighted its untapped potential in regulating mood, stress, and sleep via neurotransmitter production.

Several bacterial strains, including lactic acid bacteria, bifidobacteria and others, have demonstrated GABA production capabilities. However, the magnitude of GABA output varies among these strains, and their efficacy in GABA synthesis within the human gastrointestinal environment is uncertain. This stems from the fact that GABA synthesis, typically a pH-stress response, stalls in less acidic environments.

Lactiplantibacillus plantarum Lp815 stands out. Using advanced computational and high-throughput screening techniques, we identified this strain's superior GABA production capability. Remarkably, it synthesizes a significant amount of GABA within the physiologically relevant pH range.

The study will evaluate self-reported sleep disturbance in a broad age-range of adults who have chosen to try this product. The study will incorporate participant reported outcome questionnaires and surveys, the use of a health tracking wearable device to explore objective digital outcome measures of sleep, heart rate and heart rate variability and in a subset of participants, the study will utilize an at-home urinary test to evaluate neurotransmitter levels in the body. There is no "doctor-patient" relationship as part of this research since the participant as a consumer is making the informed choice to take the product and take part in the observational process with self-reported measures and a simple urine test that can be done at home. Findings from this study will contribute knowledge toward the dosing and formulation of the probiotic product and the design of future studies.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Has self-reported sleep disturbance
* Insomnia Severity Index (ISI) score of > 15, with score on question on difficulty falling asleep > 2 ("moderate") at screening
* Interested in understanding more about their sleep and choose to use the probiotic product
* Willing to do a 1-week washout out of any OTC or other products for sleep and/or (e.g. melatonin, anticholinergics, valerian root etc.) prior to randomization and refrain from use for the duration of the study
* Willing to do a 4-week washout from any systemic antibiotic, prebiotic, probiotic and postbiotic use prior to randomization
* If taking prescription medications for sleep and/or anxiety (e.g. Benzodiazepines, zolpidem, zaleplon, SSRIs, Buspirone, Tricyclics, MAOIs), or other class of medication for sleep, must be on a "stable dose" for at least 4 weeks prior to randomization. "Stable dose" is defined as no changes in dosage or frequency of the specified medications for at least 4 weeks prior to randomization and throughout the study period.
* If using any cannabis-containing products, must be on a stable dose for at least 4 weeks prior to randomization and consume < 10 mg/day of THC
* If regularly consuming alcohol, must be willing to stay on a stable amount throughout the study period and to log alcohol consumption.
* In good general health at the time of screening (Investigator discretion).
* Able to read and understand English.
* Able to read, understand, and provide informed consent.
* Able to use a personal smartphone device and download Chloe by People Science.
* Able to receive shipment of the product at an address within the United States.
* Is willing to wear, sync daily, and charge twice weekly a provisioned health tracking wearable device (Oura ring) everyday (up to 7 weeks) during sleep. If the participant already has an Oura ring, they can use their own device and account.
* Able to complete study assessments over the course of up to 7 weeks.

Exclusion Criteria:

* Do not have a smartphone and/or internet access.
* Concomitant Therapies:

  * Participants taking prescription medication for sleep and/or anxiety (e.g. Benzodiazepines, zolpidem, zaleplon, SSRIs, Buspirone, Tricyclics, MAOIs) not on a stable dose for at least 4 weeks
  * Participants receiving Cognitive Behavioral Therapy for Insomnia (CBTi)
  * Participants receiving any investigational therapies or treatments within 30 days prior to randomization.
  * Participants taking any other prescription medications that impact systemic GABA levels (e.g., GABA supplements, barbiturates, gabapentin, pregabalin, valproate, tiagabine, vigabatrin, baclofen)
  * Participants currently taking or have taken probiotics, prebiotics or postbiotics within the past 4 weeks prior to randomization.
  * Current antibiotic use or use within 4 weeks prior to randomization.
* Other Illnesses or Conditions: Participants who have the following conditions or comorbidities are excluded:

  * Confirmed diagnoses of the following sleep disorders: Narcolepsy, Restless Leg Syndrome, Circadian Rhythm Disorders
  * Confirmed diagnosis of Sleep Apnea that is untreated or not well controlled
  * Known diagnosis of Inflammatory Bowel Disease (Crohn's Disease or Ulcerative Colitis) or Irritable Bowel Syndrome
  * Current or prior history of psychotic disorder
  * Confirmed diagnosis of major depressive disorder or bipolar disorder
  * Diagnosed with Alcohol or Substance Abuse Disorder
  * Currently pregnant, planning to become pregnant in the next 1 month, or breastfeeding
  * Presence of any infection or illness that causes chronic night-waking or impairs ability to retain urine overnight (e.g., chronic pain, uncontrolled benign prostatic hyperplasia, prostatitis, urinary tract infection, catheterization, etc.).
  * Have a significant illness, disease or condition which, in the opinion of the principal investigator, may impact their ability to participate in the trial or impact the trial outcomes.
* Known hypersensitivity or previous allergic reaction to microcrystalline cellulose (MCC).
* Presence of another environmental factor that severely impacts sleep quality (e.g., a new baby, pet or other loved one that wakes frequently or needs frequent care or feeding throughout the night)
* Work in an environment requiring shift work (e.g., rotating shifts, night shifts, or irregular hours).
* Have any known and planned international travel during the study period.
* Are unlikely for any reason to be able to comply with the trial or considered unsuited for participation in the study by the Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Generally healthy participants (all genders) 18 years or older who have self-reported sleep disturbance with a score of >15 on the screening Insomnia Severity Index questionnaire.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Observe differences in sleep outcomes | Participants will complete up to a 16-week study consisting of screening period, randomization and shipping period, a baseline period, and a 6-week product/placebo use period.
  The primary outcome is to observe differences in sleep outcomes between the GABA Probiotic and the placebo control group from intake and baseline to the end of the study period.
  This will be measured by a change in the Insomnia Sleep Index (ISI) score between placebo and study product group. Baseline period will be compared as well. On a scale of 0-28, a higher score indicates more severe insomnia, which is a worse outcome.

SECONDARY OUTCOMES:
Evaluate the impact of GABA Probiotic on anxiety | Participants will complete up to a 16-week study consisting of screening period, randomization and shipping period, a baseline period, and a 6-week product/placebo use period.
  A secondary outcome is to evaluate the impact of GABA Probiotic on anxiety.
  This will be measured by a change in Generalized Anxiety Disorder-7 (GAD-7) score between placebo and study product group. Baseline period will be compared as well. On a scale between 0-21, a higher Generalized Anxiety Disorder score indicates more severe anxiety, which is a worse outcome.
Evaluate the impact of GABA Probiotic on gastrointestinal symptoms | Participants will complete up to a 16-week study consisting of screening period, randomization and shipping period, a baseline period, and a 6-week product/placebo use period.
  A secondary outcome is to evaluate the impact of GABA Probiotic on gastrointestinal symptoms.
  This will be measured by a change in Gastrointestinal Symptom Rating Scale (GSRS) score between placebo and study product group. Baseline period will be compared as well. The Gastrointestinal Symptom Rating Scale uses a 7-point Likert scale, where 1 means no discomfort and 7 means severe discomfort. A higher score indicates more severe gastrointestinal symptoms, which is a worse outcome.
Evaluate the impact of GABA Probiotic on subjective sleep quality | Participants will complete up to a 16-week study consisting of screening period, randomization and shipping period, a baseline period, and a 6-week product/placebo use period.
  A secondary outcome is to evaluate the impact of GABA Probiotic on subjective sleep quality.
  This will be measured by a change in average sleep quality score as measured by daily 10-point visual analogue rating scale (VAS) between placebo and study product group. Baseline period will be compared as well. A higher score between 0-10, will indicate poor sleep quality and a worse outcome.
Evaluate the impact of GABA Probiotic on daytime alertness | Participants will complete up to a 16-week study consisting of screening period, randomization and shipping period, a baseline period, and a 6-week product/placebo use period.
  A secondary outcome is to evaluate the impact of GABA Probiotic on daytime alertness.
  This will be measured by a change in average daytime alertness score between placebo and study product group as measured by a daily 10-point VAS scale. Baseline period will be compared as well. A higher score between 0-10, will indicate better sleep quality and a better outcome.
Evaluate the impact of GABA Probiotic on mood | Participants will complete up to a 16-week study consisting of screening period, randomization and shipping period, a baseline period, and a 6-week product/placebo use period.
  A secondary outcome is to evaluate the impact of GABA Probiotic on mood.
  This will be measured by a change in average mood score between placebo and study product group as measured by a daily 10-point VAS scale. Baseline period will be compared as well. A higher score between 0-10, will indicate better mood and a better outcome.
Evaluate the impact of GABA Probiotic on night sweats | Participants will complete up to a 16-week study consisting of screening period, randomization and shipping period, a baseline period, and a 6-week product/placebo use period.
  A secondary outcome is to evaluate the impact of GABA Probiotic on night sweats.
  This will be measured by a change in average severity score of night sweats between placebo and study product group as measured by a daily 10-point VAS scale. Baseline period will be compared as well. A higher score between 0-10, will indicate severe sweating and a worse outcome.
Evaluate the impact of GABA Probiotic on quality of life | Participants will complete up to a 16-week study consisting of screening period, randomization and shipping period, a baseline period, and a 6-week product/placebo use period.
  A secondary outcome is to evaluate the impact of GABA Probiotic on quality of life.
  This will be measured by a change in average quality of life score between placebo and study product group as measured by a daily 10-point VAS scale. Baseline period will be compared as well. A higher score between 0-10, will indicate better quality of life and a better outcome.
Evaluate the impact of GABA Probiotic on improvement in sleep | Participants will complete up to a 16-week study consisting of screening period, randomization and shipping period, a baseline period, and a 6-week product/placebo use period.
  A secondary outcome is to evaluate the impact of GABA Probiotic on participants' overall subjective impression of improvement in sleep.
  This will be measured by a change from baseline in Patient Global Impression of Change (P-GIC) score between placebo and study product group. On a scale between 1-7, a higher score means greater improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Noah Craft, MD, Principal Investigator — People Science, Inc.
Locations (1):
- People Science, Inc., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan currently to share IPD with other researchers.

REFERENCES:
- [Derived] Grant AD, Erfe MCB, Delebecque CJ, Keller D, Zimmerman NP, Kazaryan A, Oliver PL, Moos J, Luna V, Craft N. Lactiplantibacillus plantarum Lp815 improves sleep and increases urinary GABA in a randomized, double-blind, placebo-controlled study of sleep disturbance. Sci Rep. 2026 Jan 19;16(1):644. doi: 10.1038/s41598-025-27861-6. PMID 41554764